CLINICAL TRIAL: NCT02628301
Title: Is Microvascular Dysfunction an Early Phenomenon in the Development of Skeletal Muscle Insulin Resistance? A Dietary Intervention Study in Healthy Men
Brief Title: Microvascular Dysfunction and the Development of Whole-body Insulin Resistance
Acronym: DESIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erik Serne, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DC2014DES001
Record Dates: First submitted 2015-03-10; First posted 2015-12-11 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Insulin Resistance; Type 2 Diabetes; Obesity
Keywords: Obesity; Type 2 Diabetes Mellitus; Hypercaloric diet; Microcirculation; Microvascular dysfunction; Insulin Resistance; Insulin Sensitivity; Insulin signaling
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypercaloric diet (Active Comparator): Hypercaloric diet (1.6x REE) for 30 days
  Interventions: Dietary Supplement: Hypercaloric diet
- Normal diet (Placebo Comparator): Normocaloric diet (1.0xREE)
  Interventions: Other: Normocaloric diet

INTERVENTIONS:
Dietary Supplement: Hypercaloric diet — Hypercaloric diet consisting of 60% excess calories based on resting energy expenditure (REE). Calories will be provided in the form of snacks in between the ad libitum meals. A subsequent hypocaloric diet will consist of 1.0x resting energy expenditure.
  Arms: Hypercaloric diet
Other: Normocaloric diet — Normocaloric diet
  Arms: Normal diet

SUMMARY:
This study aims to elucidate the role of the microcirculation in the development of whole body insulin resistance. The investigators hypothesize that impaired insulin signaling in the vasculature is an early phenomenon in the development of whole body insulin resistance. Furthermore, the investigators aim to identify improvement of microvascular function as a potential target in diabetes prevention and treatment.

DETAILED DESCRIPTION:
In today's society, food availability grossly exceeds our body's caloric demands. Excessive caloric intake causes weight gain and induces insulin resistance, a common characteristic of obesity and major risk factor for type 2 diabetes (T2DM) and cardiovascular disease.

The primary targets of insulin action are skeletal muscle, adipose tissue and the liver, but recent data point to the vascular endothelium as an important target. Insulin directly targets the endothelial cell where it activates phosphoinositide 3-kinase, resulting in Akt-mediated phosphorylation of endothelial nitric oxide synthase (eNOS). This leads to NO production - a potent vasodilator in the human body. Simultaneously insulin also activates the mitogen-activated protein kinase pathway in endothelial cells, which enhances the generation of the vasoconstrictor endothelin-1 via extracellular signal-regulated kinases 1/2 signaling. Via these two pathways insulin can regulate vascular tone.

In healthy individuals, insulin signaling in the endothelial cell leads to capillary recruitment in skeletal muscle tissue via vasodilatation of terminal arterioles. It has been proposed that insulin in this matter regulates the delivery of insulin and glucose to skeletal muscle by increasing endothelial surface area. In obese individuals and patients with T2DM, insulin-mediated capillary recruitment in skeletal muscle tissue is impaired and insulin-dependent glucose uptake is diminished. Whether these two processes are linked or occur in parallel remains unknown.

Interestingly, studies in rodents demonstrated that during obesity induced by high fat feeding, insulin resistance develops in the vasculature before these responses are detected in muscle, liver, or adipose tissue. Therefore, insulin signaling in endothelium might change in response to a positive energy balance to prevent nutrient overload in muscle and optimize nutrient storage in adipose tissue. Conversely, it has been hypothesized that early reversal of endothelial insulin resistance could prevent peripheral insulin resistance, assuming a cause-and-effect relationship between these processes. The most compelling evidence for this hypothesis came from studies in endothelial cell specific insulin receptor substrate-2 (IRS-2) knock-out mice. Kubota et al. demonstrated that impaired insulin signaling in endothelial cells, due to reduced IRS-2 expression and insulin-induced eNOS phosphorylation, caused attenuation of insulin-induced capillary recruitment and insulin delivery, which reduced glucose uptake by skeletal muscle. Moreover, restoration of insulin-induced eNOS phosphorylation in endothelial cells by infusion of beraprost sodium - a stable prostaglandin analogue - completely reversed the reduction in capillary recruitment and insulin delivery in tissue-specific knockout mice lacking IRS-2 in endothelial cells and fed a high-fat diet. As a result, glucose uptake by skeletal muscle was restored in these mice.

These data suggest that pharmacological stimulation of tissue perfusion may hold promise as a therapeutic strategy to increase whole body glucose disposal and thus prevent or reduce hyperglycaemia. In humans however, data linking improvement of capillary recruitment by pharmacological agents to restoration of whole-body glucose uptake are lacking. Low dose iloprost infusion - another stable prostaglandin analogue - has been shown to improve insulin-stimulated whole-body glucose uptake, but the mechanistic role of microvascular response was not assessed. Overall, it remains to be demonstrated whether improving capillary recruitment by endothelial insulin signaling or direct stimulation of smooth muscle tissue may serve as an attractive preventive or therapeutic approach to bypass cellular resistance to glucose disposal.

In conclusion, vascular insulin resistance leads to blunted capillary recruitment in the skeletal muscle and may lead to diminished glucose uptake due to a decreased capillary surface area for nutrient exchange. Up till now however it remains unclear if these processes are interrelated or occur in parallel. Evidence from animal studies suggest that vascular insulin resistance precedes diminished whole-body glucose uptake and myocellular impairments. This indicates a potential cause-effect relationship. In humans, however, this was never demonstrated. On the other hand, decreased capillary recruitment of skeletal muscle tissue could also protect muscle tissue from nutrient overload and shunt excess calories towards adipose tissue. Presently, it is unknown whether insulin redistributes blood flow from skeletal muscle to adipose tissue during hypercaloric conditions. Finally, it is unknown if stimulation of tissue perfusion with a pharmacological agent can restore whole-body glucose uptake is therefore an effective strategy in prevention or treatment of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* BMI 22-25 kg/m2
* Normal insulin sensitivity as estimated by Homeostasis Model Assessment (HOMA-IR)
* Normoglycemia as defined by fasting plasma glucose (FPG) <6.1 mmol/l
* Normoglycemia as defined by 2 h glucose <7.8 mmol/l during oral glucose tolerance test (OGTT)
* Normal diet pattern according to the Dutch guidelines for a healthy diet 2006
* Stable body weight (<3% weight change) during 6 months before enrolment in the study

Exclusion Criteria:

* Presence of any relevant disease
* Use of any relevant medication
* First-degree relative with type 2 diabetes
* Smoking
* Shift work
* A history of chronic glucocorticoids (GC) use or GC use < 3 months ago
* Excessive sport activities (more often than 3 hours per week)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Microvascular Insulin Sensitivity | Baseline, 7-10 days after initiation of the hypercaloric diet, after the hypercaloric diet, after the subsequent hypocaloric diet
  Capillary recruitment by contrast-enhanced ultrasound.

SECONDARY OUTCOMES:
Whole Body Insulin Sensitivity | Baseline, 7-10 days after initiation of the hypercaloric diet, after the hypercaloric diet,
  M-value by euglycemic-hyperinsulinemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Erik Serne, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saltiel AR, Kahn CR. Insulin signalling and the regulation of glucose and lipid metabolism. Nature. 2001 Dec 13;414(6865):799-806. doi: 10.1038/414799a. PMID 11742412
- [Background] Kim JA, Montagnani M, Koh KK, Quon MJ. Reciprocal relationships between insulin resistance and endothelial dysfunction: molecular and pathophysiological mechanisms. Circulation. 2006 Apr 18;113(15):1888-904. doi: 10.1161/CIRCULATIONAHA.105.563213. PMID 16618833
- [Background] De Boer MP, Meijer RI, Wijnstok NJ, Jonk AM, Houben AJ, Stehouwer CD, Smulders YM, Eringa EC, Serne EH. Microvascular dysfunction: a potential mechanism in the pathogenesis of obesity-associated insulin resistance and hypertension. Microcirculation. 2012 Jan;19(1):5-18. doi: 10.1111/j.1549-8719.2011.00130.x. PMID 21883642
- [Background] Kim F, Pham M, Maloney E, Rizzo NO, Morton GJ, Wisse BE, Kirk EA, Chait A, Schwartz MW. Vascular inflammation, insulin resistance, and reduced nitric oxide production precede the onset of peripheral insulin resistance. Arterioscler Thromb Vasc Biol. 2008 Nov;28(11):1982-8. doi: 10.1161/ATVBAHA.108.169722. Epub 2008 Sep 4. PMID 18772497
- [Background] Barrett EJ, Eggleston EM, Inyard AC, Wang H, Li G, Chai W, Liu Z. The vascular actions of insulin control its delivery to muscle and regulate the rate-limiting step in skeletal muscle insulin action. Diabetologia. 2009 May;52(5):752-64. doi: 10.1007/s00125-009-1313-z. Epub 2009 Mar 13. PMID 19283361
- [Background] Park SY, Cho YR, Kim HJ, Higashimori T, Danton C, Lee MK, Dey A, Rothermel B, Kim YB, Kalinowski A, Russell KS, Kim JK. Unraveling the temporal pattern of diet-induced insulin resistance in individual organs and cardiac dysfunction in C57BL/6 mice. Diabetes. 2005 Dec;54(12):3530-40. doi: 10.2337/diabetes.54.12.3530. PMID 16306372
- [Background] Kubota T, Kubota N, Kumagai H, Yamaguchi S, Kozono H, Takahashi T, Inoue M, Itoh S, Takamoto I, Sasako T, Kumagai K, Kawai T, Hashimoto S, Kobayashi T, Sato M, Tokuyama K, Nishimura S, Tsunoda M, Ide T, Murakami K, Yamazaki T, Ezaki O, Kawamura K, Masuda H, Moroi M, Sugi K, Oike Y, Shimokawa H, Yanagihara N, Tsutsui M, Terauchi Y, Tobe K, Nagai R, Kamata K, Inoue K, Kodama T, Ueki K, Kadowaki T. Impaired insulin signaling in endothelial cells reduces insulin-induced glucose uptake by skeletal muscle. Cell Metab. 2011 Mar 2;13(3):294-307. doi: 10.1016/j.cmet.2011.01.018. PMID 21356519
- [Background] Paolisso G, Di Maro G, D'Amore A, Passariello N, Gambardella A, Varricchio M, D'Onofrio F. Low-dose iloprost infusion improves insulin action in aged healthy subjects and NIDDM patients. Diabetes Care. 1995 Feb;18(2):200-5. doi: 10.2337/diacare.18.2.200. PMID 7537193
- [Derived] Emanuel AL, Meijer RI, Woerdeman J, van Raalte DH, Diamant M, Kramer MHH, Serlie MJ, Eringa EC, Serne EH. Effects of a Hypercaloric and Hypocaloric Diet on Insulin-Induced Microvascular Recruitment, Glucose Uptake, and Lipolysis in Healthy Lean Men. Arterioscler Thromb Vasc Biol. 2020 Jul;40(7):1695-1704. doi: 10.1161/ATVBAHA.120.314129. Epub 2020 May 14. PMID 32404008